CLINICAL TRIAL: NCT05289908
Title: Phase I/II Clinical Trial of Intrathecal Pemetrexed as First Line Intrathecal Chemotherapy in Patients With Leptomeningeal Metastasis
Brief Title: Intrathecal Pemetrexed for Leptomeningeal Metastasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Affiliated Hospital of Guangdong Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guangdong 999 Brain Hospital (Other); The Second Hospital of Hebei Medical University (Other); Panjin Liaoyou Gem Flower Hospital (Unknown); Wuxi People's Hospital (Other); Huizhou Third People's Hospital, Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, The First Hospital of Jilin University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PMLM
Record Dates: First submitted 2022-03-10; First posted 2022-03-22 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-11

CONDITIONS: Leptomeningeal Metastases
Keywords: Leptomeningeal metastasis; Intrathecal chemotherapy; Pemetrexed
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Pemetrexed; Folic Acid; Vitamin B 12; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase I study (Experimental): Pemetrexed (Alimta, Eli Lilly and Company) is administrated by intrathecal injection, plus dexamethasone 5 mg, twice per week for 2 weeks, followed by once per week for 4 weeks. The initial dose of intrathecal pemetrexed is 15 mg, escalated to 20 mg, and then 25 mg.... A minimum of three patients and a maximum of six are enrolled in each cohort. Folic acid 200-400 μg is administered orally once daily, prior to the first intrathecal pemetrexed, until 21 days after the last intrathecal pemetrexed. A single dose of vitamin B12 1000 μg is administered by intramuscular injection before the first intrathecal pemetrexed, once per 3 weeks.
  Interventions: Drug: Pemetrexed (1); Drug: Folic Acid; Drug: Vitamin B12; Drug: Dexamethasone
- Phase II study (Experimental): Pemetrexed (Alimta, Eli Lilly and Company) is administrated by intrathecal injection, plus dexamethasone 5 mg, twice per week for 2 weeks, followed by once per week for 4 weeks. The maximum-tolerated dose determined in phase I study is chosen as the treatment dose in phase II study.
  Interventions: Drug: Pemetrexed (2); Drug: Folic Acid; Drug: Vitamin B12; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pemetrexed (1) — Pemetrexed (Alimta, Eli Lilly and Company) is administrated by intrathecal injection, plus dexamethasone, twice per week for 2 weeks, followed by once per week for 4 weeks. The initial dose of intrathecal pemetrexed is 15 mg, escalated to 20 mg, and then 25 mg....
  Arms: Phase I study
Drug: Pemetrexed (2) — The maximum-tolerated dose determined in phase I study is chosen as the treatment dose in phase II study.
  Arms: Phase II study
Drug: Folic Acid — Folic acid 200-400 μg is administered orally once daily, prior to the first intrathecal pemetrexed, until 21 days after the last intrathecal pemetrexed.
Drug: Vitamin B12 — A single dose of vitamin B12 1000 μg is administered by intramuscular injection before the first intrathecal pemetrexed, once per 3 weeks.
Drug: Dexamethasone — Dexamethasone, 5 mg, intrathecal injection via lumbar puncture, simultaneously with pemetrexed, twice per week for 2 weeks, followed by once per week for 2-4 weeks.

SUMMARY:
Intrathecal chemotherapy is one of the most important treatment modalities for leptomeningeal metastasis of solid tumors. In the previous study(Intrathecal Pemetrexed for Recurrent Leptomeningeal Metastasis From Non-small Cell Lung Cancer: A Prospective Pilot Clinical Trial. ClinicalTrials.gov identification number: NCT03101579), pemetrexed presented feasibility of intrathecal administration. Pemetrexed at 10 mg dose level on the schedule of 1-2 times per week was recommended as an intrathecal administration agent for patients with refractory leptomeningeal metastases from non-small-cell lung cancer in the previous study. Moreover, the maximum-tolerated dose and recommended dose of intrathecal pemetrexed in the previous study was obtained without vitamin supplementation. Vitamin supplementation has been shown to reduce pemetrexed-induced myelosuppression. In this study, the regimen of intrathecal pemetrexed with folic acid and vitamin B12 supplementation may provide higher safety. Therefore, the purpose of this study is to investigate the maximally tolerated dose and evaluate the safety and effectiveness of intrathecal pemetrexed with vitamin supplementation as the first-line intrathecal chemotherapy in patients with leptomeningeal metastases from malignant solid tumors.

DETAILED DESCRIPTION:
This is a phase I/II clinical trial. The objective of the study is patients with leptomeningeal metastases from solid tumors. Pemetrexed (Alimta, Eli Lilly and Company) is administrated by intrathecal injection, plus dexamethasone 5 mg, twice per week for 2 weeks, followed by once per week for 4 weeks. In phase I study, the initial dose of intrathecal pemetrexed is 15 mg, escalated to 20 mg, and then 25 mg.... A minimum of three patients and a maximum of six are enrolled in each cohort. A dose-limiting toxicity is defined as grade 3 neurological toxicities (e.g., chemical meningitis) or other grade 4 toxicity. If none of the three patients experiences any dose-limiting toxicity, the subsequent three patients are enrolled at the next higher dosage level. If one of three patients experiences a dose-limiting toxicity, up to three more patients are enrolled at the same level. The maximum-tolerated dose is defined as the dose where 0/3 or 1/6 patients experiences a dose-limiting toxicity with at least two patients encountering dose-limiting toxicity at the higher dose. If more than two patients experience a dose-limiting toxicity, that level is considered too toxic. The maximum-tolerated dose is exceeded and an additional three patients should be treated at the next lower dose level. Folic acid 200-400 μg is administered orally once daily, prior to the first intrathecal pemetrexed, until 21 days after the last intrathecal pemetrexed. A single dose of vitamin B12 1000 μg is administered by intramuscular injection before the first intrathecal pemetrexed, once per 3 weeks. In phase II study, the maximum-tolerated dose determined in phase I study is chosen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been definitely diagnosed as leptomeningeal metastasis according to cerebrospinal fluid cytology or neuroimaging, or patients who got the clinical diagnosis by combining with the history of cancer, clinical manifestation, cerebrospinal fluid examination, neuroimaging etc.;
2. Patients who have been diagnosed as malignant solid tumor according histopathology or cytopathology combined with imaging;
3. No prior intrathecal chemotherapy;
4. Normal liver and kidney function; WBC≥4000/mm3, Plt≥100000/mm3;
5. No other severe chronic diseases;
6. No history of severe nervous system disease;
7. No severe dyscrasia.

Exclusion Criteria:

1. Patients receiving molecularly targeted drugs that are effective in treating leptomeningeal metastases within 2 weeks prior to enrollment;
2. Patients with hydrocephalus or other factors suggestive of cerebrospinal fluid circulation obstruction;
3. patients with serious central nervous system disorders including severe encephalopathy, moderate or severe coma, and Glasgow Coma Score of <8 points;
4. Patients who have been diagnosed as hematological malignancy or primary central germ cell tumor;
5. Other reasons that were unsuitable for this study, including patients with lethal or extensive systemic diseases with few treatment options,psychiatric illness and poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose | From the beginning of the treatment until two months after the treatment.
  A dose-limiting toxicity (DLT) was defined as grade 3 neurological toxicities (e.g. chemical meningitis) or other grade 4 toxicity. If more than two patients experienced a DLT, that level was considered too toxic. The maximal tolerated dose (MTD) was exceeded and an additional three patients should be treated at the next lower dose level. The MTD was defined as the dose where 0/3 or 1/6 patients experienced a DLT with at least two patients encountering DLT at the higher dose.
Incidence of treatment-related adverse events | From the beginning of the treatment until two months after the treatment.
  The incidence of treatment-related adverse events were measured for determining tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03). Events of grade 3-5 are defined as moderate and severe adverse events.

SECONDARY OUTCOMES:
Overall survival time | The evaluation was performed at least 7 months after leptomeningeal metastasis diagnosis or until death.
  Survival time was defined from the enrollment until death or the last follow-up.

OTHER OUTCOMES:
Clinical response rate | From the beginning of the treatment until two months after the treatment or when patient died.
  The Response Assessment in Neuro-Oncology (RANO) criteria proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be available to other researchers.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.
Access Criteria: Individual participant data will be public accessable via contacting with principal investigator by email within 6 months after the trial complete.

REFERENCES:
- [Background] Pan Z, Yang G, He H, Cui J, Li W, Yuan T, Chen K, Jiang T, Gao P, Sun Y, Cong X, Li Z, Wang Y, Pang X, Song Y, Zhao G. Intrathecal pemetrexed combined with involved-field radiotherapy as a first-line intra-CSF therapy for leptomeningeal metastases from solid tumors: a phase I/II study. Ther Adv Med Oncol. 2020 Jul 17;12:1758835920937953. doi: 10.1177/1758835920937953. eCollection 2020. PMID 32733606
- [Background] Pan Z, Yang G, Cui J, Li W, Li Y, Gao P, Jiang T, Sun Y, Dong L, Song Y, Zhao G. A Pilot Phase 1 Study of Intrathecal Pemetrexed for Refractory Leptomeningeal Metastases From Non-small-cell Lung Cancer. Front Oncol. 2019 Aug 30;9:838. doi: 10.3389/fonc.2019.00838. eCollection 2019. PMID 31544065
- [Derived] Pan Z, Ye X, Huang Y, Tai P, Liu M, Sun X, Tang R, Gu A, Wang Z, Shen L, Pang X, Yuan T, Yang G. Intrathecal pemetrexed for newly diagnosed leptomeningeal metastases: a multicenter, open-label, phase I/II study. J Neurooncol. 2025 Nov;175(2):857-868. doi: 10.1007/s11060-025-05160-4. Epub 2025 Jul 23. PMID 40699526